CLINICAL TRIAL: NCT04142086
Title: Safety, Tolerability, and Immunogenicity Dose-ranging Study of the Investigational Yellow Fever Vacine (vYF) Candidate Vaccine in Adults
Brief Title: Dose-ranging Study of an Investigational Yellow Fever Candidate Vaccine in Adults
Acronym: VYF01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VYF01; U1111-1217-1958 (Other: UTN)
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Yellow Fever (Healthy Volunteers)
MeSH Terms: conditions — Yellow Fever | interventions — Yellow Fever Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An observer-blind procedure is followed for the injection of vYF or YF-VAX. Neither the observer Investigator, nor the Sponsor, nor the participants know product is administered. The "vaccinator" is in charge of preparing and administering the products and is not authorized to collect any safety data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Experimental): 1 injection of vYF vaccine Dosage 1
  Interventions: Biological: Yellow fever vaccine (produced on serum-free Vero cells), Dosage 1 vYF vaccine
- Group 2 (Experimental): 1 injection of vYF vaccine Dosage 2
  Interventions: Biological: Yellow fever vaccine (produced on serum-free Vero cells), Dosage 2 vYF vaccine
- Group 3 (Experimental): 1 injection of vYF vaccine Dosage 3
  Interventions: Biological: Yellow fever vaccine (produced on serum-free Vero cells), Dosage 3 vYF vaccine
- Group 4 (Active Comparator): 1 injection of YF-VAX
  Interventions: Biological: Yellow fever vaccine

INTERVENTIONS:
Biological: Yellow fever vaccine (produced on serum-free Vero cells), Dosage 1 vYF vaccine — Pharmaceutical form: Powder and diluent for suspension for injection Route of administration: Subcutaneous
  Arms: Group 1
Biological: Yellow fever vaccine (produced on serum-free Vero cells), Dosage 2 vYF vaccine — Pharmaceutical form: Powder and diluent for suspension for injection Route of administration: Subcutaneous
  Arms: Group 2
Biological: Yellow fever vaccine (produced on serum-free Vero cells), Dosage 3 vYF vaccine — Pharmaceutical form: Powder and diluent for suspension for injection Route of administration: Subcutaneous
  Arms: Group 3
Biological: Yellow fever vaccine — Pharmaceutical form: Powder and diluent for suspension for injection Route of administration: Subcutaneous
  Other Names: YF-VAX
  Arms: Group 4

SUMMARY:
The primary objectives of the study are:

* To describe the safety profile of each of the 3 dosages of vYF and of YF-VAX® within the 28 days post-vaccination and up to the 6 months (Day 180) post-vaccination visit
* To describe the antibody responses elicited by each of the 3 dosages of vYF and by YF-VAX on Day 0 pre-vaccination and then on Day 10, Day 14, Day 28 and 6 months (Day 180) post-vaccination overall and by baseline flavivirus serostatus
* To quantify the detectable yellow fever (YF) vaccinal viremia in each vaccine groups (vYF and YF-VAX) in a subset of subjects on Day 0 visit, Day 1 visit, Day 3 visit, Day 5 visit, Day 7 visit, Day 10 visit, and Day 14 visit.

DETAILED DESCRIPTION:
Study duration per participant is approximately 6 months.

ELIGIBILITY:
Inclusion criteria :

* Aged 18 years up to 60 years on the day of inclusion
* Able to read and understand the Informed Consent Form which has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures

Exclusion criteria:

* Participant is pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination. To be considered of non-childbearing potential, a female must be pre-menarche , or post-menopausal for at least 1 year, or surgically sterile
* Participation at the time of study enrollment (or in the 4 weeks preceding the trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine in the 4 weeks following the trial vaccination
* Previous vaccination against a flavivirus disease including YF with either the trial vaccine or another vaccine
* Receipt of immune globulins, blood, or blood-derived products in the past 6 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy, or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known history of flavivirus infection
* Known systemic hypersensitivity to any of the vaccine components, eggs, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances
* Known history or laboratory evidence of human immunodeficiency virus infection
* Known history of hepatitis B or hepatitis C seropositivity
* Personal of family history of thymic pathology (thymoma, thymectomy, or myasthenia)
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion, including malignancy, such as leukemia or lymphoma
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 100.4 F). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Administration of any anti-viral within 2 months preceding the vaccination and up to the 6 weeks following the vaccination
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study
* Planned travel in a YF endemic country within 6 months of investigational or control vaccine administration

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with immediate adverse events | Within 30 minutes after vaccination
  Immediate adverse events are any unsolicited systemic adverse events reported in the 30 minutes after vaccination
Number of participants with solicited injection site reactions | Within 7 days after vaccination
  Solicited injection site reactions include injection site pain, erythema and swelling
Number of participants with solicited systemic reactions | Within 14 days after vaccination
  Solicited systemic reactions include fever, headache, malaise, and myalgia
Number of participants with unsolicited adverse events | Within 28 days after vaccination
  Unsolicited (spontaneously reported) adverse events not fulfilling criteria for solicited adverse reactions
Number of participants with Grade 3 fever | Within 28 days after vaccination
  Grade 3 fever is defined as temperature ≥ 102.1°F
Number of participants with serious adverse events | From Day 0 to Day 180
  Serious adverse events are collected throughout the study
Number of participants with hematology and biochemistry out-of-range test results | From Day 0 to Day 14
  Hematology and biochemistry values that are out-of-range are assessed
Number of participants with YF and flavivirus viremia and out-of-normal-range biological test results in the event of severe fever, or suspicion of neurotropic disease or acute viscerotropic diseases | Within 28 days after vaccination
  Investigators are provided with guidelines for recognition and assessment of potential viscerotropic and neurotropic events
Number of participants with seroconversion to YF virus | From Day 0 to Day 28
  Seroconversion is defined as a fourfold increase in neutralizing antibody titers as compared to pre-vaccination value. Seroconversion is assessed from Day 0 (pre-vaccination) to Day 10, Day 14 and Day 28.
Number of participants with neutralizing antibody titers against YF virus above pre-defined threshold | From Day 0 to Day 180
  Pre-defined threshold of 10 1/dilution
Geometric mean titers of neutralizing antibodies against YF virus | From Day 0 to Day 180
  Geometric mean titer ratio Day 10/Day 0, Day 14/Day 0, Day 28/Day 0 and Day 180/Day 0
Number of participants with YF vaccinal viremia | From Day 0 to Day 14
  Vaccinal viremia is measured by YF specific quantitative reverse transcription polymerase chain reaction (RT-PCR) assay in samples collected on Day 0, Day 1, Day 3, Day 5, Day 7, Day 10, and Day 14.
Level of YF vaccinal viremia | From Day 0 to Day 14
  Vaccinal viremia is measured by YF specific quantitative RT-PCR assay in samples collected on Day 0, Day 1, Day 3, Day 5, Day 7, Day 10, and Day 14.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Investigational Site Number 8400001, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Pagnon A, Carre C, Aguirre M, Chautard E, Gimenez S, Raynal F, Feroldi E, Scott P, Modjarrad K, Vangelisti M, Mantel N. Next generation yellow fever vaccine induces an equivalent immune and transcriptomic profile to the current vaccine: observations from a phase I randomised clinical trial. EBioMedicine. 2024 Oct;108:105332. doi: 10.1016/j.ebiom.2024.105332. Epub 2024 Sep 17. PMID 39293214
- See also: VYF01 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25385&tenant=MT_SNY_9011